CLINICAL TRIAL: NCT06636136
Title: Transtibial Osseointegration Surgery Study (TOSS)
Brief Title: Transtibial Osseointegration
Acronym: TOSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2023-0445
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Amputation; Traumatic, Leg, Lower
Keywords: Transtibial; Osseointegration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- OPRA implant leg (Other): The participants will have two stage surgical procedures to implant the OPRA device to the amputated leg.
  Interventions: Device: OPRA

INTERVENTIONS:
Device: OPRA — Surgery

SUMMARY:
Purpose:

Aim 1: Quantify soft tissue complications and infections of service members with transtibial amputations treated with OPRA OI and compare them to transfemoral OI service members.

Aim 2: Compare the validated domains, such as functional, quality of life and pain scores, from the preoperative baseline to follow-up visits to determine if persons with transtibial amputations treated with OPRA osseointegrated prostheses demonstrate statistically significant and clinically relevant improvements.

Aim 3: Compare physical performance measures preoperatively to follow-up visits for persons with transtibial amputations treated with OPRA osseointegrated prostheses to quantify statistically significant and clinically relevant improvements.

Aim 4: Quantify the biomechanical loading and bone quality changes that are directly associated with patient reported outcomes for persons with transtibial amputations treated with OPRA osseointegration.

Aim 5: Compare outcome measures between persons with traditional socket prostheses (patients as self-controls) and OPRA OI devices as well as a comparison between persons with transtibial OI and transfemoral OI.

Subject Population:

Male and female military health care beneficiaries age 22 to 65 years old presenting with a Transtibial limb loss.

Study Design:

This is a 4-year, prospective cohort FDA pivotal study involving off-label use of the OPRA OI implant in persons with transtibial amputation.

Procedures:

SURGICAL PROCEDURES:

Surgery Stage I:

The distal part of the tibia is exposed, preferably using existing incisions, to produce an appropriate fasciocutaneous flap. By the use of fluoroscopy and guiding devices the correct position of the fixture in the medullary canal is found. The canal is reamed step by step to a proper diameter to facilitate insertion of the implant. If the bone quality is poor, as determined by the operating surgeon, autologous bone graft from the iliac crest and/or the medullary canal is used. The fixture is then implanted into the intramedullary canal. Careful surgical technique is essential not to damage the tissue and to achieve osseointegration. A central screw, healing cylinder, and healing bolt are inserted. A myodesis is performed, and the wound is closed using suture.

The sutures are removed 2-3 weeks postoperatively. When the skin is completely healed the Patient's conventional socket prosthesis could, in some instances, be used.

Surgery Stage II (3-5 months after Stage I):

The tibia is exposed via the incision from the Stage I-Surgery. The healing cylinder is removed and the tissues are trimmed in a way that the distal end of the bone protrudes a few millimeters. The skin will be attached directly to it. The endosteal canal is reamed to facilitate placement of the abutment. The skin in the abutment area is then trimmed to a diameter equal to the protruding end of the tibia. This is done to remove the subcutaneous fat and facilitate healing of the dermal layer to the distal end of the bone. The subcutaneous tissue is affixed to the periosteum using absorbable suture to prevent skin movement. A 8mm punch biopsy tool is used to create a circular hole in the skin precisely over the residual tibial canal. The remaining portion of the fasciocutaneous flap is sutured into position. A bolster dressing is placed and routine postoperative wound care is performed by daily dressing changes. Sutures are removed 2-3 weeks postoperatively.

CLINICAL PROCEDURES

A pre-study visit will be conducted up to 6 months prior to Surgery Stage I. Postoperative visits will occur 2-3 weeks after each surgery. Additional follow-up visits will occur 6, 12, 24, 36, 48 and 60 months post-Surgery Stage II. It is standard of care to follow patients postoperatively from time to time to ensure the wound(s) is /are healing, surveil for complications, and ensure rehabilitation is progressing. That said, the sole reason for engaging in the Clinical Follow-Up Procedures is for the purpose of conducting research under this particular protocol. Additional visits may occur including x-rays at the discretion of the clinical investigator in order to monitor the participants medical status/bone healing.

RESEARCH PROCEDURES

Timepoints: Baseline, Post-Op Stage II, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months

The patients will be assessed before and after the surgery regularly. Both performance and safety data will be recorded on specially designed electronic Case Report Forms (eCRFs). Clinical and radiological assessments are performed preoperatively (in connection with the surgical procedures.

DETAILED DESCRIPTION:
The patients will be regularly assessed during the follow-up period after the surgery. Both performance and safety data will be recorded on specially designed electronic Case Report Forms (eCRFs). Clinical and radiological assessments are performed preoperatively (in connection with the surgical procedures) and at 6, 12, 24, 36, 48 and 60 months (after completion of the surgical treatment).

Prior to surgery the participant will have had their completed skeletal growth verified by radiographs and/or CT scans.

The participants will be asked to refrain from taking NSAID and salicylates for two weeks prior to and 6 weeks after surgery.

Procedures will be performed by the study PI and AI, Drs. Potter and Anderson, respectively. Each has considerable experience in the treatment of combat related limb loss, and the surgical procedures necessary to implant the OPRA device.

SUMMARY OF THE SURGICAL PROCEDURES Surgery Stage I The distal part of the tibia is exposed, preferably using existing amputation incisions, to produce an appropriate fasciocutaneous flap. Under fluoroscopic guidance, the canal is reamed step by step to a proper diameter to facilitate insertion of the implant. The fixture is then implanted into the intramedullary canal under fluoroscopic guidance. Careful surgical technique is essential not to damage the tissue and to achieve osseointegration. A central screw, healing cylinder, and healing bolt are inserted. A myoplasty is performed, and the wound is closed using sutures.

Surgery Stage II (3-6 months after Stage I) Through a limited incision, the graft screw and components are removed. Then cutaneous flaps are elevated and muscle is trimmed and then the muscle fascia is attached to the bone approximately 1.5cm proximal to the distal tibia using 0-vicryl. A purse string stitch is then used to further reinforce the myoplasty. The cutaneous flap is thinned and identified a suitable position for the skin penetration aperture on the superior flap. A 8mm punch biopsy tool is used to create the aperture. Using the abutment as a guide, the fat layer is removed to expose the undersurface of the dermis. A drain is placed exiting proximally on the lateral or medial side. The flap is then rotated and fixed into position using a series of 2-0 Vicryl stutures. The Abutment is then inserted and the threads were cleaned with an angiocatheter and saline flush. The abutment screw is tightened by hand. The anterior flap is then trimmed for closure and the incision is closed with 2-0 Monocryl, 3-0 Monocryl and a self-adhering mesh with 2-octyl cyanoacrylate liquid adhesive. Nitropaste is placed around the aperture and an antimicrobial foam dressing bolster. This is held in place using the skate-board wheel (donut) provided for this purpose. The patient remains on bedrest for 5 days to allow healing of the aperture site and skin flaps.

CLININCAL PROCEDURES A pre-study visit will be conducted up to 6 months prior to Surgery Stage I. Postoperative visits will occur 2-3 weeks after each surgery. Additional follow-up visits will occur 6, 12, 24, 36, 48, and 60 months post-Surgery Stage II. It is standard of care to follow patients postoperatively from time to time to ensure the wound(s) is /are healing, surveil for complications, and ensure rehabilitation is progressing. That said, the sole reason for engaging in the Clinical Follow-Up Procedures is for the purpose of conducting research under this particular protocol. Additional visits may occur including x-rays at the discretion of the clinical investigator in order to monitor the participants medical status/bone healing status.

X-ray, CT scan and function performance measure procedures are standard care. RESEARCH PROCEDURES Timepoints: Baseline, Post-Op Stage II, 6 months, 12 months, 24 months, 36 months, 48 months and 60 months.

The participants will have up to 7 postoperative visits after each surgery.

All questionnaires and DEXA are being administered / performed for research purpose. The DEXA scans will be performed at the Department of the Physical Medicine and Rehabilitation in the Biomechanics Lab at WRNMMC.

Baseline Collection Patient Demographic characteristics, amputation demographic characteristics, Medication list. Questionnaires: Q-TFA, OPUS (functional status, health quality of life index, satisfaction of device and service and Clinical Survey), PROMIS (Physical Functions, Pain Interference and Pain Behavior), EQ-5D, DVPRS, Tampa Scale for Kinesiophobia (TSK), Functional Performance: DEXA, Physical Mobility:Time Up and Go (TUG), Four Square Step Test (4SST), 6-Minute Walk Test, Amputee Mobility Predictor (AMP), Comprehensive High-Level Activity Mobility Predictor (CHAMP), Bilateral Amputee Mobility Predictor (BAMP) (for bilateral amputee only), 5 Time Sit to Stand (5TSTS), and Metabolic Energy Expenditure and Radiography: X-ray and CT Scan.

Post-Op Stage II Surgery Questionnaires: Q-TFA, OPUS (functional status, health quality of life index and satisfaction of device and service), PROMIS (Physical Functions, Pain Interference and Pain Behavior), EQ-5D, DVPRS, Medication List, and Tampa Scale for Kinesiophobia (TSK) and Radiography: X-rays.

6 Months Questionnaires: Q-TFA, OPUS (functional status, health quality of life index and satisfaction of device and service), PROMIS (Physical Functions, Pain Interference and Pain Behavior), EQ-5D, DVPRS, Medication List, Tampa Scale for Kinesiophobia (TSK),and Radiography: X-rays.

12 Months Questionnaires: Q-TFA, OPUS (functional status, health quality of life index, and satisfaction of device and service), PROMIS (Physical Functions, Pain Interference and Pain Behavior), EQ-5D, DVPRS, Medication List, Tampa Scale for Kinesiophobia (TSK), Functional Performance: DEXA, Physical Mobility (Time Up and Go (TUG), Four Square Step Test (4SST), 6-Minute Walk Test, Amputee Mobility Predictor (AMP), Comprehensive High-Level Activity Mobility Predictor (CHAMP), Bilateral Amputee Mobility Predictor(BAMP)(for bilateral amputees only), 5 Time Sit to Stand (5TSTS), and Metabolic Energy Expenditure and Radiography: X-rays.

24 Months Questionnaires: Q-TFA, OPUS (functional status, health quality of life index, satisfaction of device and service and Clinical Survey), PROMIS (Physical Functions, Pain Interference and Pain Behavior), EQ-5D, DVPRS, Medication List, Tampa Scale for Kinesiophobia (TSK), Functional Performance: DEXA, Physical Mobility Time Up and Go (TUG), Four Square Step Test (4SST), 6-Minute Walk Test, Amputee Mobility Predictor (AMP), Comprehensive High-Level Activity Mobility Predictor (CHAMP), Bilateral Amputee Mobility Predictor (BAMP)(for bilateral amputees only), 5 Time Sit to Stand (5TSTS), and Metabolic Energy Expenditure and Radiography: X-rays.

36 Months Questionnaires: Q-TFA, OPUS (functional status, health quality of life index, satisfaction of device and service and Clinical Survey), PROMIS (Physical Functions, Pain Interference and Pain Behavior), EQ-5D, DVPRS, Medication List, Tampa Scale for Kinesiophobia (TSK), Functional Performance: DEXA, Physical Mobility Time Up and Go (TUG), Four Square Step Test (4SST), 6-Minute Walk Test, Amputee Mobility Predictor (AMP), Comprehensive High-Level Activity Mobility Predictor (CHAMP), Bilateral Amputee Mobility Predictor (BAMP)(for bilateral amputees only), 5 Time Sit to Stand (5TSTS), and Metabolic Energy Expenditure and Radiography: X-rays.

48 Months Questionnaires: Q-TFA, OPUS (functional status, health quality of life index, satisfaction of device and service and Clinical Survey), PROMIS (Physical Functions, Pain Interference and Pain Behavior), EQ-5D, DVPRS, Medication List, Tampa Scale for Kinesiophobia (TSK), Functional Performance: DEXA, Physical Mobility Time Up and Go (TUG), Four Square Step Test (4SST), 6-Minute Walk Test, Amputee Mobility Predictor (AMP), Comprehensive High-Level Activity Mobility Predictor (CHAMP), Bilateral Amputee Mobility Predictor (BAMP)(for bilateral amputees only), 5 Time Sit to Stand (5TSTS), and Metabolic Energy Expenditure and Radiography: X-rays.

60 Months Questionnaires: Q-TFA, OPUS (functional status, health quality of life index, satisfaction of device and service and Clinical Survey), PROMIS (Physical Functions, Pain Interference and Pain Behavior), EQ-5D, DVPRS, Medication List, Tampa Scale for Kinesiophobia (TSK), and Decision Regret, Functional Performance: DEXA, Physical Mobility Time Up and Go (TUG), Four Square Step Test (4SST), 6-Minute Walk Test, Amputee Mobility Predictor (AMP), Comprehensive High-Level Activity Mobility Predictor (CHAMP), Bilateral Amputee Mobility Predictor (BAMP)(for bilateral amputees only), 5 Time Sit to Stand (5TSTS), and Metabolic Energy Expenditure and Radiography: X-rays.

QUESTIONNAIRES Q-TFA (Questionnaire for Persons with a Transfemoral Amputation) A disease specific questionnaire evaluating functional and HRQL in limb loss population.

OPUS-The Orthotic and Prosthetic User's Survey is a self-report questionnaire used for quality assessment, to maintain awareness of improvement activities, to evaluate changes in patient's functional status and quality of life and assess satisfaction with devices and services (functional status, health quality of life index, satisfaction of device and service and Clinical Survey).

PROMIS Patient-Reported Outcomes Measurement Information System. Physical Function: Measures the outcome of patients with musculoskeletal disorders by assessing physical function through a grading scale of activities of daily living.

Pain Interference: Measures the extent to which pain hinders an individual's engagement with physical, mental, cognitive, emotional, recreational, and social activities.

Pain Behavior: Measure self-reported external manifestations of pain. EQ-5D a valid and reliable family of questionnaires to measure of health-related quality of life. If the participant's answers indicate they may be depressed, they will be referred to behavioral health for further assessment.

DVPRS a pain assessment tool that utilizes a numerical rating scale enhanced by functional word descriptors, color coding, and pictorial facial expressions matched to pain levels.

Medication List Listing the medication the participant is taking. Tampa Scale for Kinesiophobia (TSK) a 17-item questionnaire that quantifies fear of movement.

Sane Score a single-question outcome measure that asks patients to rate their function, as it pertains to the area being treated, on a scale of 0 to 100.

Decision Regret a question asking the participant if they would have the surgery again.

FUNTIONAL PERFORMANCE Timed up and Go (TUG) a measure of physical mobility. Four Square Step Test (4SST) an objective reliable measure of dynamic balance that assesses the ability to step over objects forward, sideways and backward.

6-Minute Walk Test (6MWT) an objective measure of mobility. Amputee Mobility Predictor (AMP) provides a tool for measuring ambulation potential and can be administered either with or without prosthesis.

Comprehensive High-Level Activity Mobility Predictor (CHAMP) a performance-based assessment used to measure higher level of functional mobility, and consists of four advanced physical tests (single-limb stance test, Edgren side step test, T-test, and Illinois agility test).

Bilateral Amputee Mobility Predictor (BAMP) the AMP for bilateral amputees' biomechanical outcomes derived from gait evaluation.

5 Time Sit to Stand (5TSTS) a test used to assess instructed to stand up from sitting for five minutes as quickly as possible without using the hands for support.

Metabolic Energy Expenditure Breath-by-breath oxygen consumption and heart rate will be measured continuously during a 5-10-minute rest, followed by walking trail(s) at multiple speeds with each of sufficient length to achieve steady-state.

DEXA Whole body composition will be measured using linear fan beam dual energy x-ray absorptiometry. Whole body composition scans will be performed on up to 4 localized sites (5 sites for those with bilateral TF limb loss); spine (L1-L4), bilateral Femur neck (hip), and "Gruen zones" (around the osseointegrated implant).

10.2 Data Collection: Describe all the data variables, information to be collected, the source of the data, and how the data will be operationally measured.

A study team member will collect information on our source documentation from the study participant or through participant's medical records at the following time points: Baseline/screening, 2-3 week post-operative from surgery stage II, 6 months, 12 months, 24 months, 36 months, 48 months and 60 months.(from surgery stage II). Data will be entered into REDCap.

Baseline (collected from the participant at initial screening) Eligibility Checklist Patient Demographics Characteristics Amputation Demographic Characteristics Medication list Questionnaires Q-TFA OPUS Functional Status Quality of life of Life Index Satisfaction of Device and Services Clinical Survey PROMIS Physical Function Pain Interference Pain Behavior EQ-5D DVPRS Medication List Tampa Scale for Kinesiophobia (TSK) Clinical Assessment ** Physical Exam Pregnancy Test ( if applicable) Functional Performance DEXA TUG 4SST 6-Minute Walk Test AMP CHAMP Bilateral Amputee Mobility Predictor* 5TSTS Metabolic Energy Expenditure Radiography** X-rays CT Post-Op Surgery Stage II Questionnaires Q-TFA OPUS Functional Status Quality of life of Life Index Satisfaction of Device and Services PROMIS Physical Function Pain Interference Pain Behavior EQ-5D DVPRS Medication List Tampa Scale for Kinesiophobia (TSK) Radiography** X-rays Clinical Assessment** Date of assessment, skin penetration area assessment; normal conditions, redness, secretion, superficial infections, deep infection, infection history, physical exam, adverse event assessment

6 Months Follow Up Questionnaires Q-TFA OPUS Functional Status Quality of life of Life Index Satisfaction of Device and Services PROMIS Physical Function Pain Interference Pain Behavior EQ-5D DVPRS Medication List Tampa Scale for Kinesiophobia (TSK) Radiography** X-rays Clinical Assessment** Date of assessment, skin penetration area assessment; normal conditions, redness, secretion, superficial infections, deep infection, infection history, physical exam, adverse event assessment

12 Months Follow Up Questionnaires Q-TFA OPUS Functional Status Quality of life of Life Index Satisfaction of Device and Services Clinical Survey PROMIS Physical Function Pain Interference Pain Behavior EQ-5D DVPRS Medication List Tampa Scale for Kinesiophobia (TSK) Functional Performance DEXA TUG 4SST 6-Minute Walk Test AMP CHAMP Bilateral Amputee Mobility Predictor* 5TSTS Metabolic Energy Expenditure Radiography** X-rays Clinical Assessment** Date of assessment, skin penetration area assessment; normal conditions, redness, secretion, superficial infections, deep infection, infection history, physical exam, adverse event assessment.

24 Months Follow Up Questionnaires Q-TFA OPUS Functional Status Quality of life of Life Index Satisfaction of Device and Services Clinical Survey PROMIS Physical Function Pain Interference Pain Behavior EQ-5D DVPRS Medication List Tampa Scale for Kinesiophobia (TSK) Functional Performance DEXA TUG 4SST 6-Minute Walk Test AMP CHAMP Bilateral Amputee Mobility Predictor* 5TSTS Metabolic Energy Expenditure Radiography** X-rays Clinical Assessment** Date of assessment, skin penetration area assessment; normal conditions, redness, secretion, superficial infections, deep infection, infection history, physical exam, adverse event assessment.

36 Months Follow Up Questionnaires Q-TFA OPUS Functional Status Quality of life of Life Index Satisfaction of Device and Services Clinical Survey PROMIS Physical Function Pain Interference Pain Behavior EQ-5D DVPRS Medication List Tampa Scale for Kinesiophobia (TSK) Functional Performance DEXA TUG 4SST 6-Minute Walk Test AMP CHAMP Bilateral Amputee Mobility Predictor* 5TSTS Metabolic Energy Expenditure Radiography** X-rays Clinical Assessment** Date of assessment, skin penetration area assessment; normal conditions, redness, secretion, superficial infections, deep infection, infection history, physical exam, adverse event assessment.

48 Months Follow Up Questionnaires Q-TFA OPUS Functional Status Quality of life of Life Index Satisfaction of Device and Services Clinical Survey PROMIS Physical Function Pain Interference Pain Behavior EQ-5D DVPRS Medication List Tampa Scale for Kinesiophobia (TSK) Functional Performance DEXA TUG 4SST 6-Minute Walk Test AMP CHAMP Bilateral Amputee Mobility Predictor* 5TSTS Metabolic Energy Expenditure Radiography** X-rays Clinical Assessment** Date of assessment, skin penetration area assessment; normal conditions, redness, secretion, superficial infections, deep infection, infection history, physical exam, adverse event assessment.

60 Months Follow Up Questionnaires Q-TFA OPUS Functional Status Quality of life of Life Index Satisfaction of Device and Services Clinical Survey PROMIS Physical Function Pain Interference Pain Behavior EQ-5D DVPRS Medication List Tampa Scale for Kinesiophobia (TSK) Decision Regret Functional Performance DEXA TUG 4SST 6-Minute Walk Test AMP CHAMP Bilateral Amputee Mobility Predictor* 5TSTS Metabolic Energy Expenditure Radiography** X-rays Clinical Assessment** Date of assessment, skin penetration area assessment; normal conditions, redness, secretion, superficial infections, deep infection, infection history, physical exam, adverse event assessment.

* For bilateral amputees only

** For clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a transtibial amputation age 22-65.
* The OPRA™ Implant System is indicated for patients who have transtibial amputation due to trauma or cancer and who have or are anticipated to have rehabilitation problems with, or cannot use, a conventional socket prosthesis. The OPRA™ Implant System is intended for skeletally mature patients.
* The patient failed to receive benefit from socket prostheses or is expected to not tolerate socket use due to problems such as:

  * Recurrent skin infections and ulcerations in the socket contact area
  * Pain
  * A short stump preventing the use of socket prosthesis
  * Volume fluctuation in the stump
  * Soft tissue scarring
  * Extensive area of skin grafting
  * Socket retention problems due to excessive perspiration
  * Restricted mobility
* Eligible to receive care at Military Treatment Facility
* DEERS-eligible

Exclusion Criteria:

* The patient's skeletal growth is not complete. Completed skeletal growth is defined through the finding of generally closed epiphyseal zones on X-ray.
* The patient has atypical skeletal anatomy which may affect treatment with OPRA™.

  * Examples of atypical skeletal anatomy.
  * Skeletal dimensions outside defined interval.
  * Development anomalies.
  * Conditions which are not amenable to device insertion such as deformities, fracture, infection.
* The patient would have less than 2 mm of remaining cortex bone available around the implant, if implanted.
* Osteoporosis.
* The patient is older than 65 years and younger than 22 years.
* BMI over 35.
* Do not treat patients with the following concurrent diseases:

  * Severe peripheral vascular disease.
  * Diabetic mellitus with complications.
  * Neuropathy or neuropathic disease.
  * Active infection or dormant bacteria.
  * Metabolic bone disease and/or metastatic lesions in the residual tibia.
* Pregnancy before the surgery female patients will take a pregnancy test) Note: Patients who become pregnant, after surgery stage I, surgery stage II will be delayed until safe to do so by their doctor. The patient will remain in the study, unless they would like to withdrawal.
* The patient is not expected to be able to comply with treatment and follow up requirements.
* Participants unable to sign their own consent (No legally authorized representatives may provide consent)

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Quantify soft tissue complications of participants with transtibial amputations treated with OPRA OI and compare them to transfemoral OI service participants | 60 months post-surgery stage II.
  Collecting the rate of complications after the surgery
Compare the validated domains: functional from the preoperative baseline to follow-up visits | 60 months post-surgery stage II.
  The participants reported outcome measurement system: Questionnaire
  · To evaluate "before and after surgery" changes in functional status
Quantify soft tissue infections of participants with transtibial amputations treated with OPRA OI and compare them to transfemoral OI service participants | 60 months post-surgery stage II.
  Collecting the rate of infections after the surgery
Compare the validated domains: quality of life from the preoperative baseline to follow-up visits | 60 months post-surgery stage II.
  The participants reported outcome measurement system: Questionnaire
  · To evaluate "before and after surgery" changes in quality of life
Compare the validated domains: pain scores from the preoperative baseline to follow-up visits | 60 months post-surgery stage II.
  The participants reported outcome measurement system: Questionnaire
  · To evaluate "before and after surgery" changes in pain

SECONDARY OUTCOMES:
Compare physical performance measures ( changes in residual limb confidence ) preoperatively to follow-up visits for persons within transtibial amputations treated with OPRA osseointegrated prostheses | 60 months post-surgery stage II.
  · To evaluate "before and after surgery" changes in residual limb confidence (or kinesiophobia)
Quantify the biomechanical loading changes that are directly associated with patient-reported outcomes for persons with transtibial amputations treated with OPRA osseointegration. | 60 months post-surgery stage II.
  · To evaluate "before and after surgery" changes in gait biomechanics; provides an objective measure(s) for evaluating the quality of movement during walking.
  6-Minute Walk Test (a measure of mobility)
Compare outcome measures between persons with traditional socket prostheses (patients as self-controls) and OPRA OI devices as well as a comparison between persons with transtibial OI and transfemoral OI. | 60 months post-surgery stage II.
  * Quantify the differences in outcome measures and biomechanical performance between persons with traditional socket prostheses and persons with OI devices.
    * Amputee Mobility Predictor (AMP) (as a measure of ambulation potential)
    * Bilateral Amputee Mobility Predictor (BAMP) (If the participants are bilateral amputees, they will have this procedure done)
  * Compare the outcome measures and biomechanical performance of persons with transfemoral OI and transtibial OI.
    * Amputee Mobility Predictor (AMP) (as a measure of ambulation potential)
    * Bilateral Amputee Mobility Predictor (BAMP) (If the participants are bilateral amputees, they will have this procedure done)
Compare physical performance measures (in functional muscle strength) preoperatively to follow-up visits for persons within transtibial amputations treated with OPRA osseointegrated prostheses to quantify statistically significant and clinically relevant | 60 months post-surgery stage II.
  To evaluate "before and after surgery" changes in functional muscle strength:
Compare physical performance measures (changes in physical mobility) preoperatively to follow-up visits for persons within transtibial amputations treated with OPRA osseointegrated prostheses | 60 months post-surgery stage II.
  · To evaluate "before and after surgery" changes in physical mobility
Compare physical performance measures (changes in body composition ) preoperatively to follow-up visits for persons within transtibial amputations treated with OPRA osseointegrated prostheses | 60 months post-surgery stage II.
  · To evaluate "before and after surgery" changes in body composition:
Compare physical performance measures ( changes in metabolic energy expenditure) preoperatively to follow-up visits for persons within transtibial amputations treated with OPRA osseointegrated prostheses | 60 months post-surgery stage II.
  · To evaluate "before and after surgery" changes in metabolic energy expenditure.
Quantify bone quality changes that are directly associated with patient-reported outcomes for persons with transtibial amputations treated with OPRA osseointegration. | 60 months post-surgery stage II.
  · To evaluate "before and after surgery" changes in bone mineral density
  DEXA- whole body composition will be measured using linear fan beam dual-energy x-ray absorptiometry. Whole body composition scans will be performed on up to 4 localized sites (5 sites for those with bilateral TF limb loss); spine (L1-L4), bilateral Femur neck (hip), and "Gruen zones" (around the osseointegrated implant)

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Tintle, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (2):
- United States (2):
  - Orhopaedic Surgery Service, Walter Reed National Military Medical Center, Bethesda, Maryland
  - Department of Orthopaedic Surgery and Department of Anesthesiology & Critical Care Penn Medicine University City, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Adell R, Lekholm U, Rockler B, Branemark PI. A 15-year study of osseointegrated implants in the treatment of the edentulous jaw. Int J Oral Surg. 1981 Dec;10(6):387-416. doi: 10.1016/s0300-9785(81)80077-4. PMID 6809663
- [Result] Adell R, Eriksson B, Lekholm U, Branemark PI, Jemt T. Long-term follow-up study of osseointegrated implants in the treatment of totally edentulous jaws. Int J Oral Maxillofac Implants. 1990 Winter;5(4):347-59. PMID 2094653
- [Result] Hakansson B, Carlsson P. Skull simulator for direct bone conduction hearing devices. Scand Audiol. 1989;18(2):91-8. doi: 10.3109/01050398909070728. PMID 2756338
- [Result] Li Y, Lindeque B. Percutaneous Osseointegrated Prostheses for Transfemoral Amputations. Orthopedics. 2018 Mar 1;41(2):75-80. doi: 10.3928/01477447-20180227-03. PMID 29566253
- [Result] Zaid MB, O'Donnell RJ, Potter BK, Forsberg JA. Orthopaedic Osseointegration: State of the Art. J Am Acad Orthop Surg. 2019 Nov 15;27(22):e977-e985. doi: 10.5435/JAAOS-D-19-00016. PMID 31181031
- [Result] Hagberg K. Bone-anchored prostheses in patients with traumatic bilateral transfemoral amputations: rehabilitation description and outcome in 12 cases treated with the OPRA implant system. Disabil Rehabil Assist Technol. 2019 May;14(4):346-353. doi: 10.1080/17483107.2018.1449016. Epub 2018 Mar 14. PMID 29534624
- [Result] Branemark R, Berlin O, Hagberg K, Bergh P, Gunterberg B, Rydevik B. A novel osseointegrated percutaneous prosthetic system for the treatment of patients with transfemoral amputation: A prospective study of 51 patients. Bone Joint J. 2014 Jan;96-B(1):106-13. doi: 10.1302/0301-620X.96B1.31905. PMID 24395320
- [Result] Morris CD, Potter BK, Athanasian EA, Lewis VO. Extremity amputations: principles, techniques, and recent advances. Instr Course Lect. 2015;64:105-17. PMID 25745899
- [Result] Harness N, Pinzur MS. Health related quality of life in patients with dysvascular transtibial amputation. Clin Orthop Relat Res. 2001 Feb;(383):204-7. doi: 10.1097/00003086-200102000-00023. PMID 11210955
- [Result] Leijendekkers RA, van Hinte G, Frolke JP, van de Meent H, Atsma F, Nijhuis-van der Sanden MW, Hoogeboom TJ. Functional performance and safety of bone-anchored prostheses in persons with a transfemoral or transtibial amputation: a prospective one-year follow-up cohort study. Clin Rehabil. 2019 Mar;33(3):450-464. doi: 10.1177/0269215518815215. Epub 2018 Dec 12. PMID 30537856
- [Result] Atallah R, Li JJ, Lu W, Leijendekkers R, Frolke JP, Al Muderis M. Osseointegrated Transtibial Implants in Patients with Peripheral Vascular Disease: A Multicenter Case Series of 5 Patients with 1-Year Follow-up. J Bone Joint Surg Am. 2017 Sep 20;99(18):1516-1523. doi: 10.2106/JBJS.16.01295. PMID 28926380
- [Result] Akhtar MA, Hoellwarth JS, Al-Jawazneh S, Lu W, Roberts C, Al Muderis M. Transtibial Osseointegration for Patients with Peripheral Vascular Disease: A Case Series of 6 Patients with Minimum 3-Year Follow-up. JB JS Open Access. 2021 Jun 23;6(2):e20.00113. doi: 10.2106/JBJS.OA.20.00113. eCollection 2021 Apr-Jun. PMID 34235362
- [Result] Hagberg K, Branemark R, Hagg O. Questionnaire for Persons with a Transfemoral Amputation (Q-TFA): initial validity and reliability of a new outcome measure. J Rehabil Res Dev. 2004 Sep;41(5):695-706. PMID 15558399
- [Result] McGlothlin AE, Lewis RJ. Minimal clinically important difference: defining what really matters to patients. JAMA. 2014 Oct 1;312(13):1342-3. doi: 10.1001/jama.2014.13128. No abstract available. PMID 25268441
- [Result] Wright A, Hannon J, Hegedus EJ, Kavchak AE. Clinimetrics corner: a closer look at the minimal clinically important difference (MCID). J Man Manip Ther. 2012 Aug;20(3):160-6. doi: 10.1179/2042618612Y.0000000001. PMID 23904756
- [Result] Hung M, Saltzman CL, Kendall R, Bounsanga J, Voss MW, Lawrence B, Spiker R, Brodke D. What Are the MCIDs for PROMIS, NDI, and ODI Instruments Among Patients With Spinal Conditions? Clin Orthop Relat Res. 2018 Oct;476(10):2027-2036. doi: 10.1097/CORR.0000000000000419. PMID 30179950